CLINICAL TRIAL: NCT00374010
Title: Improving Patient-clinician Communication Among End-stage Renal Disease African Patients and Their Families
Brief Title: Improving Patient-clinician Communication About End-of-life Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0412044
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2008-03

CONDITIONS: End-stage Renal Disease
Keywords: end-of-life decision making; advance care planning
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Patient-Centered Advance Care Planning — The PC-ACP is a scheduled interview with the dyad, delivered by a trained nurse facilitator. It consists of 5 stages and lasts about an hour:
  1. Representational assessment (10 - 15 minutes);
  2. Exploring concerns related to planning for future medical decision-making (10 - 15 minutes);
  3. Creating conditions for conceptual change (5 minutes);
  4. Introducing replacement information using a disease-specific Statement of Treatment Preferences document (15 minutes); and
  5. Summary (3 - 5 minutes)

SUMMARY:
The specific aims are:

1. to evaluate the feasibility and acceptability of PC-ACP among African American patients with End-stage Renal Disease and their surrogates and
2. to examine preliminary effects of PC-ACP on patient and surrogate outcomes (patients' perceived quality of communication, surrogates' level of comfort in decision making for the patient, patients' difficulty in making choices, patient-surrogate congruence in goals of care, and patients' and surrogates' psychosocial/spiritual receptiveness) at one week following receipt of the intervention.

DETAILED DESCRIPTION:
Despite the increasing emphasis placed on patient-clinician communication about end of life care, efforts to guide the patient to make an informed end-of-life treatment decision often fail. Past efforts to enhance end-of-life discussions were insufficient to create treatment decisions that were consistent with the patient's values and the surrogate's ability to make end-of-life decisions for his/her loved one when required. The importance of effective end-of-life discussions has been documented extensively, yet systematic explorations of the effects of such dialogue with African Americans are nearly absent from the literature. The proposed study is designed to test the ability of an hour-long intervention, Patient-Centered Advance Care Planning (PC-ACP), to enhance clinicians' communication about end-of-life care with patients and surrogates. The specific aims are (1) to evaluate the feasibility and acceptability of PC-ACP among African American patients with End-stage Renal Disease and their surrogates and (2) to examine preliminary effects of PC-ACP on patient and surrogate outcomes (patients' perceived quality of communication, surrogates' level of comfort in decision making for the patient, patients' difficulty in making choices, patient-surrogate congruence in goals of care, and patients' and surrogates' psychosocial/spiritual receptiveness) at one week following receipt of the intervention. A randomized, controlled, pre and post study will be conducted. Subjects (patient-surrogate dyads) will be randomized to PC-ACP or to a usual care control group. Data to assess feasibility, clinical and sociodemographic data, and baseline measures of patient and surrogate outcomes will be collected when subjects enter the study. Measures of the patient and surrogate outcomes and data to assess acceptability of the intervention will be administered at one week follow up. Findings from this study are critical to strengthening PC-ACP and designing a randomized controlled trial to test its efficacy for improving the quality of patient-clinician communication and the quality of decision making for future medical care with African American patients, in comparison with non-Hispanic Whites.

ELIGIBILITY:
Inclusion Criteria:

1. have been on either center-hemodialysis or home-peritoneal dialysis
2. are cognitively intact,i.e., able to communicate, able to understand information, able to make choices and give rationale,
3. have an individual who can be present during the intervention as a surrogate decision maker,
4. are over 18 years of age, and
5. are able to communicate in English. Surrogates must be over 18 years of age and be able to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-01; Primary Completion 2007-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
congruence between patient and surrogate at one week after intervention | one week post intervention
patient and surrogate satisfaction with communication | one week post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Kyung Song, PhD, Principal Investigator — University of Pittsburgh School of Nursing